CLINICAL TRIAL: NCT05425680
Title: Clinical Effectiveness and Biomechanics Study for Remote Intelligent Interactive Virtual Reality Assessment and Rehabilitation in Patients With Degenerative Lumbar Spine Diseases
Brief Title: Remote Intelligent Interactive Virtual Reality Assessment in Patients With Degenerative Lumbar Spine Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202201047RINC
Record Dates: First submitted 2022-06-13; First posted 2022-06-21 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Degenerative Lumbar Spine Diseases
Keywords: degenerative lumbar spine disease; virtual reality; telehealth; real-time detection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Core muscle training (Experimental): specific rehabilitation exercise for improving functional movements
  Interventions: Other: Core muscle training

INTERVENTIONS:
Other: Core muscle training — Combining virtual reality technology and waist wearable sensors, training the pelvis and lumbar spine movements as the main training goal, it is estimated that two 1-hour training sessions per week, a total of 6 weeks of training, to improve the core muscle of patients with lumbar degenerative diseases muscle strength.

SUMMARY:
This study will combine virtual reality (VR) technology with machine learning to focus on functional movement. Patients' symptoms will be evaluated, and exercise instruction with real-time feedback will be provided. The goals of this research are to: (1) develop a waist digital sensor for real-time monitoring as an evaluation tool, (2) apply a real-time monitoring system in conjunction with virtual reality for telerehabilitation, and (3) develop the standard model.

DETAILED DESCRIPTION:
The remote assessment and training in this study can assist patients obtaining physical therapy care at home. It is suitable for patients who avoid going to the hospital due to the epidemic, and solve the problem of long-term treatment. The outcomes will provide DLSD patients tele-rehabilitation platform and system, help medical personnel to treat patients more effectively in the future, and reduce the burden of medical costs on close ones.

ELIGIBILITY:
Inclusion Criteria:

1. able to stand and walk for 5 minutes independently
2. aged between 50 and 80 years
3. received a diagnosis of DLSD based on imaging

Exclusion Criteria:

1. neurological disorder such as stroke or spinal cord injury
2. metabolic disease such as diabetes mellitus
3. vestibular disease such as Meniere's disease.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Functional assessment: Walking speed | 6 months
  Functional assessment is a process that allows for the identification of disability. The data from the functional assessment is used to calculate walking speed (unit: m/s).
Functional assessment: Walking distance | 6 months
  Functional assessment is a process that allows for the identification of disability. The data from the functional assessment is used to calculate walking distance (unit: m).
Functional assessment: Duration | 6 months
  Functional assessment is a process that allows for the identification of disability. The data from the functional assessment is used to calculate calculate the duration it took to complete the test (unit: s).
Postural balance | 6 months
  he postural balance measurements are performed by using a inertial sensor. The data from the inertial sensor is used to calculate the 95% confidence ellipse area (unit: cm^2)
Kinematic variables: Joint angles | 6 months
  A motion capture system is used to measure the joint kinematics. The data is used to calculate joint angles (unit: degree).
Kinematic variables: Center of mass | 6 months
  A motion capture system is used to measure the displacement of the center of mass. The data is used to calculate the displacement of the center of mass (unit: cm).
Kinetic variables | 6 months
  A motion capture system is used to measure the joint kinetics. The data is used to calculate joint moments (unit: Nm)
Muscle activities | 6 months
  Electromyography is a technique for evaluating and recording muscle activity. The data from electromyography is used to calculate a normalized value (unit: ratio).

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Li Hsu, Ph.D., Principal Investigator — National Taiwan University
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital or Movement Science Lab of National Taiwan University, Taipei, Taipei
  - National Taiwan University Hospital, Taipei